CLINICAL TRIAL: NCT05593822
Title: The Relationship Between Myocardial Blush Grade and T-P-e Interval and QRS Width: Impact on In-Hospital Outcome After Successful Primary Percutaneous Coronary Intervention.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ahmed Amr Ahmed Aly, resident doctor, Assiut University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: Relationship between PPCI &ECG
Record Dates: First submitted 2022-10-09; First posted 2022-10-25 (Actual); Last update posted 2022-10-27 (Actual); Status verified 2022-10

CONDITIONS: Myocardial Infarction
MeSH Terms: conditions — Myocardial Infarction

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- patient with STEMI (Other)
  Interventions: Procedure: primary percutaneous intervention

INTERVENTIONS:
Procedure: primary percutaneous intervention — percutaneous catheterization through peripheral arteries to coronary arteries

SUMMARY:
Aim of the work:

Primary aim; is to assess relation between non invasive ECG findings, Tpe interval and QRS width and MBG in in patients with successful PCI in patients with STEMI.

Secondary aim; is to assess impact of Tpe, QRS width and MBG on in hospital outcome

DETAILED DESCRIPTION:
Primary percutaneous coronary intervention (PCI) is the treatment of choice for patients presenting with acute ST-elevation myocardial infarction (STEMI). Rapid reperfusion of infarct-related artery in STEMI is associated with substantial improvement in prognosis; however, providing epicardial flow, doesn't always mean a normal tissue perfusion. Myocardial perfusion, when assessed by myocardial blush grade (MBG) is an independent predictor of both short and long-term major adverse cardiac outcomes. (Brener SJ et al 2011, Kampinga MA 2010 and Arefin MM et al 2022)

-In this patient population, arrhythmias are also a major cause of mortality and morbidity. Repolarization heterogeneities on surface electrocardiograms (ECG) is considered as predictors of malignant ventricular arrhythmias and sudden cardiac death in patients with STEMI (Haarmark C et al 2009). The terminal part of repolarization, measured as the interval from the peak to the end of the T wave (Tpe), is a relatively indicator of risk of ventricular arrhythmias, and accumulating data suggest that T peak-to-end interval and Tpe/QT ratio are more sensitive arrhythmia markers than the older index QT dispersion (Korantzopoulos P et al 2011 Rautaharju PM et al 2005 and Duyuler PT et al 2017) ECG assessment of reperfusion therapy is mainly based on changes of the ST-segment, but the significance of the QRS duration is still not very well established. Prolonged QRS duration is associated with an increased risk of impaired ventricular systolic function and adverse effects. (Masami K et al 2011, Tsukahara K et al 2005). While ST-segment resolution is related to myocardial perfusion and cell membrane integrity, MBG reflects myocardial perfusion and microvascular patency. It is a qualitative visual assessment of the amount of contrast medium filling a territory supplied by an epicardial coronary artery. Studies are lacking that can assess the correlation between the noninvasive (QRS duration) and the invasive marker MBG of myocardial reperfusion (Yusuf J et al 2018) . The investigators will study the relation between the QRS width and MBG. The rationale was to test that whether any change in QRS duration in post-intervention patients will reflect impaired or good microvascular perfusion as assessed by the MBG.

So in the study the investigators will assess the relation between non invasive ECG findings (Tpe interval and QRS width) with invasive MBG as indicator to microvascular perfusion in patients with successful PCI in patients with STEMI and their relation to in hospital outcome

ELIGIBILITY:
Inclusion Criteria:

1. Typical ongoing ischemic chest pain for >30 minutes
2. ST elevation ≥1mm in ≥2 contiguous leads (2 mm for pericordial leads)
3. Successful primary PCI (patent infarct related artery)

Exclusion Criteria:

1. Patients with known bundle branch block
2. Patients with advanced degree of atrioventricular block or electrolyte disturbances.
3. Permanent pacemaker
4. Cardiomyopathies, chronic kidney disease.
5. Previously revascularized patients either by PCI or CABG surgery

Ages: 25 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2022-10 (Estimated); Primary Completion 2025-10 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
QRS width changes before and after PCI | 6 month
  All the patients will be suspected to the following Electrocardiogram At admission and 90 minutes after the PCI,
  -QRS complex will be measured from the start to the end of the complex,(in milli-seconds)
Tpe interval changes before and after PCI | 6 month
  All the patients will be suspected to the following Electrocardiogram At admission and 90 minutes after the PCI,
  -Tpe interval will be measured from the peak of T wave to the end of it (in milli-seconds)
MBG during PCI . | 1 year
  primary PCI The contrast density in the distal myocardial region of the IRA is graded in comparison with the blush of non-IRA myocardial regions on cine film at 25 frames per second on the best projection along at least 3 cardiac cycles duration to ensure washout.
  * Patients with no myocardial blush are graded as MBG 0,
  * those with minimal myocardial blush are graded as MBG 1,
  * those with moderate myocardial blush are graded as MBG 2
  * and patients with normal myocardial blush are graded as MBG 3.

SECONDARY OUTCOMES:
left ventricular function | 1 year
  left ventricular function before and after PCI measured by echocardiography (by simpson"s method)